CLINICAL TRIAL: NCT03904173
Title: Establishment of Molecular Profiling for Individual Clinical Routine Treatment Decision in Early Breast Cancer
Acronym: EMIT
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Klinbeforsk (Other); Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Bjørn Naume, National coordinating investigator, Oslo University Hospital
Other Study IDs: Protocol EMIT-1
Record Dates: First submitted 2019-03-06; First posted 2019-04-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Breast Neoplasms; Hormone Receptor Positive Tumor
Keywords: human epidermal growth factor receptor 2 positive; human epidermal growth factor receptor 2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed tissue, plasma, peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EMIT-1 - Multi-parameter tests: Patients with hormone sensitive HER2 negative primary breast cancer without lymph node metastasis. Treatment recommendations will be based on the Prosigna test result, in addition to conventional clinicopathological parameters.
  Interventions: Diagnostic Test: Multi-parameter tests

INTERVENTIONS:
Diagnostic Test: Multi-parameter tests — Prosigna Breast Cancer Prognostic Gene Signature Assay (PAM50) risk of recurrence (ROR) analysis CE marked assay termed Prosigna™ using digital bar code technology (NanoString Technologies Inc.).

SUMMARY:
The present project focuses on how to reduce both over- and under-treatment with adjuvant chemotherapy to a large number of breast cancer patients in Norway. A set of primary tumor prognostic factors can be analysed for potential achievement of this. Furthermore, multi-parameter tests, including detailed molecular analysis of the primary tumors might further improve the selection of patients among the lymph node negative. The study seeks to advance the development of personalised treatment of patients with early breast cancer without lymph node metastasis, by the evaluation of multi-parameter analysis as a means of identifying those patients who are likely to benefit from chemotherapy whilst sparing those who are unlikely to do so from an unnecessary and unpleasant treatment.

DETAILED DESCRIPTION:
Several known prognostic factors are used to identify breast cancer patients with an unfavourable prognosis to receive adjuvant systemic therapy, such as tumor size, histological grade, hormone receptor status and axillary lymph node metastasis. However, a large majority of early stage breast cancer patients with small primary tumors and no lymph-node metastasis receive such treatment without being at risk of developing recurrent distant disease. Furthermore, today still only about 1/3-1/2 of the patients with occult residual cancer who receive standard adjuvant chemotherapy and/or endocrine therapy are cured as a consequence of this treatment.Therefore, the future clearly needs a more precise stratification for treatment decisions. As several alternative potent therapeutic agents exist for breast cancer, a detailed characterization of the individual breast cancer disease may improve individualized prognostication and treatment. The possibilities for detailed characterization of the primary tumor have grown substantially during the last 10 years, and the prognostic and predictive impact of various molecular-based analytical tests and algorithms has been established. In order to bring forward such strategies to the individual patient in a routine clinical setting, a project with a clear goal of establishing and evaluating the most validated molecular profiles is needed.This project will evaluate the consequences of a molecular based classification of breast cancer on treatment selection as well as on economical issues such as laboratory expenses and costs related to treatment. The safety and reproducibility of the molecular assays will also be evaluated and compared to existing prognostic and predictive markers. Finally, it will also provide an opportunity for development and prospective testing of novel prognostic or predictive subtype-specific molecular markers. The project is multidisciplinary involving personnel from the following disciplines; pathology, molecular pathology, surgery, oncology and molecular biology.

Patients with lymph node negative ER+positive HER2 negative breast cancer who have completed primary surgery, are candidates for this study. Patient can be included after written informed consent has been obtained and eligibility has been established and approved. It will be organized as a multi-center study. The study will be run as a one-armed trial. Patients with appropriate primary tumor characteristics will be informed at first postoperative visit.

Treatment recommendations will be based on the Prosigna test result, in addition to conventional clinicopathological parameters. The Prosigna test will be performed after study inclusion. Before the Prosigna test result will be informed, the treating physician has to report the type of adjuvant treatment that would have been recommended without performing the Prosigna test. After the Prosigna test results is available, the final decision of adjuvant systemic treatment plan is registered.

During and after adjuvant treatment, the follow-up of patients will be according to usual care and Norwegian Breast Cancer Group (NBCG) guideline recommendations, including annual mammography and/or breast ultrasound. The events recorded during follow-up will be reported in the Norwegian Breast Cancer Registry (NBCR) which will be the main study CRF. The annual follow-up can be organized at the hospital or with the general practioner (including telephone contact from study center).

The study will recruit a total of 2150 patients, of whom approximately 1500 will not be recommended chemotherapy. After inclusion, the patients will be followed for breast cancer related events for at least 5 years (8 years from study start).

Study assessments includes the following: Demographics (age, sex) (at inclusion), medical non-breast cancer related history (not to be included in case report form, only in the medical record). Physical examination including locoregional examination of breast/chest wall and regional lymph nodes, additional examination if clinically indicated. Functional status according to NBCR.

Mammography and if indicated breast ultrasound, if not bilateral mastectomy (before surgery and at follow-up visits).Clinical status (at follow-up).

In addition to information from the patient questionnaires, patient medication (including continuation of endocrine treatment or other breast cancer treatment related medication) will be collected through the Norwegian Prescription Database and occupational disability/sick leave through the Norwegian Labor and Welfare Administration (NAV) or FD-Trygd. As the recorded patients' data in the project will be stored for a very long time, it will later be relevant to link information against the information from the Cancer Registry of Norway and the Death Cause Registry.

At baseline, 3 months, 6 months, 1 year, 2 years and at 5 year follow-up all patients will be asked to answer questionnaires consisting of established scales with good psychometric properties and single items covering socio-demographics, comorbidity, work ability, general health and quality of life (including RAND-36 and the EQ-5D), fatigue (fatigue questionnaire73), anxiety (GAD-7 questionnaire) and depressive symptoms74, life style, sleep and breast cancer specific symptoms and complaints (EORTC QLQ-BR23, FACT-B and FACT-ES).

Formal economic evaluation of cost-benefit will be performed based on simulation of treatment paths. First, an analysis of the expected cost of the interventions (patient and hospital costs) will be performed. The second step will involve an estimation of the benefits. A likely key benefit is the potential reduction in health resource use (for instance late effects that need health service and sick-leave) resulting from fewer patients treated with chemotherapy. The size of the cost/benefits will be estimated from data provided by the questionnaires as mentioned above as well as from other external sources.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (informed consent document approved by the Independent Ethics Committee [IEC]) obtained prior to any study-specific procedure
2. Female or male age ≥ 18 years
3. Able to comply with the protocol
4. Primary surgery completed or if re-resection needed, a change from pT1 to pT2 categorization is not expected
5. Histologically confirmed adenocarcinoma of the breast ≤ 5.0 cm in size (pT1-2) without metastasis to regional lymph nodes (pN0) or ≤ 20 mm in size (pT1) with lymph node micrometastases only (pN1mi)
6. Primary tumor concluded as hormone receptor positive (ER ≥ 1%), HER2 negative.

Exclusion Criteria:

1. Metastasis to regional lymph nodes or distant sites/organs.
2. Previous treatment for localized breast cancer. Previous treatment for DCIS is allowed.
3. HER2 positive
4. ER and PgR negative tumor (< 1% expression)
5. Other concomitant or earlier carcinoma less than five years prior to the breast cancer diagnosis, except for basal cell carcinoma and in situ cervix cancer
6. Use of or participation in intervention trials testing treatment with any investigational anti-cancer drug. Participation in other types of intervention trials is allowed (such participation needs to be registered).
7. Evidence of any other disease or condition that by the investigator is considered to impede follow-up of the patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary non-metastatic, node negative (pN0), hormone receptor positive, HER2 negative breast cancer. Patients with pT1pN1(mi) status may also be included.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment decision differences with or without Prosigna test | 3 years
  Differences in the number of patients receiving the various adjuvant treatments using Prosigna-test (in addition to the routine clinicopathological variables) as basis for treatment decisions compared to standard adjuvant treatment recommendations (based on clinicopathological variables only).
Distant recurrence-free interval | 8 years from study start
  Patients receiving no adjuvant chemotherapy based on Prosigna test results in combination with routine clinicopathological variables, will be recorded for metastatic events during the follow up period. To identify factors associated with survival, methods to be applied include Kaplan-Meier plots and Cox regression analyses. To statistically assess the association between breast cancer subgroups found in the analysis described above and clinical endpoints, statistical tests for comparison of survival in two or more groups (log rank test) will be used. Multivariate regression analysis will be used to adjust for other factors (such as age). Possible violations of the proportional hazards assumption inherent in both types of tests above will be detected using graphical methods as well as formal tests based on the Schoenfeld residuals.

SECONDARY OUTCOMES:
Recurrence-free interval | 8 years from study start
  Patients receiving no adjuvant chemotherapy based on Prosigna test results in combination with routine clinicopathological variables, will be recorded breast cancer recurrence events during the follow up period. To identify factors associated with survival, methods to be applied include Kaplan-Meier plots and Cox regression analyses. To statistically assess the association between breast cancer subgroups found in the analysis described above and clinical endpoints, statistical tests for comparison of survival in two or more groups (log rank test) will be used. Multivariate regression analysis will be used to adjust for other factors (such as age). Possible violations of the proportional hazards assumption inherent in both types of tests above will be detected using graphical methods as well as formal tests based on the Schoenfeld residuals.

OTHER OUTCOMES:
Patient reported outcome - EQ-5D | 3 months, 6 months, 1 year, 2 years and 5 years
  Measured by the EQ-5D questionnaire
Patient reported outcome - FACT-B/ES | 3 months, 6 months, 1 year, 2 years and 5 years
  Measured by FACT-B and FACT-ES questionnaire
Health care costs for the hospitals and society using the Prosigna test | 5 years
  To establish the cost-effectiveness (i.e. health resource use in hospitals and society) of test-directed (Prosigna) treatment strategy compared to standard practice.Formal economic evaluation of cost-benefit will be performed based on simulation of treatment paths. Firstly, an analysis of the expected cost of the interventions (patient and hospital costs) will be performed. The second step will involve an estimation of the benefits. The size of the benefits will be estimated from data provided by the clinical study as well as from other external sources. Finally, the information on costs and benefits will be used in a formal model that simulates the various treatment paths a patient can take (with the associated probabilities, costs and benefits). These simulations will lead to conclusion about the cost per quality adjusted life of the new procedures compared to the current system as well as more general social gains (including benefits such as reduced sick pay).

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Naume, MD PhD, Study Director — Oslo University Hospital
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen, Bergen
  - Drammen Hospital - Vestre Viken, Drammen, Buskerud
  - Østfold Hospital, Sarpsborg, Kalnes
  - Oslo University Hospital, Oslo, Oslo County
  - Telemark Hospital, Skien, Ulefossveien 55